CLINICAL TRIAL: NCT03747328
Title: A Phase 2a, Open-label Study to Evaluate the Safety, Tolerability, and Clinical Activity of ABI-009 (Nab-sirolimus) in Patients With Genetically-confirmed Leigh or Leigh-like Syndrome
Brief Title: ABI-009 (Nab-sirolimus) in Patients With Genetically-confirmed Leigh or Leigh-like Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND withdrawn
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS007
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Leigh Syndrome
MeSH Terms: conditions — Leigh Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABI-009 (Experimental): nanoparticle albumin bound sirolimus (ABI-009). Dose levels 1, 2.5, 5 and 10 mg/m2 given weekly for 8 cycles of ABI-009 (each cycle is weekly dosing for 2 weeks followed by a week of rest (qw2/3))
  Interventions: Drug: ABI-009

INTERVENTIONS:
Drug: ABI-009 — nanoparticle albumin bound sirolimus

SUMMARY:
A phase 2a, open-label study to evaluate the safety, tolerability, and clinical activity of ABI-009 (nab-sirolimus) in patients with genetically-confirmed Leigh or Leigh-like syndrome

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if all of the following criteria are met at screening:

1. Diagnosis of genetically-confirmed Leigh or Leigh-like syndrome, as well as documented clinical evidence (including demonstrated neurologic manifestations) of the syndrome, as confirmed by the investigator.
2. Moderate disease severity based on NPMDS score of >15 on Sections I through III, inclusive.
3. Male or female patients, ≥2 and ≤17 years of age at the time of enrollment.
4. Body weight ≥5 kg (11 lbs) at the time of enrollment.
5. Chronic, stable disease, as determined by the investigator, for a minimum of 3 months prior to enrollment. This includes, but is not limited to, patients without hospitalizations or emergency room visits, or fever <101 F, and/or acute illness.
6. Adequate liver function:

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN) mg/dL
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 x ULN.
7. Adequate renal function as defined by serum creatinine <ULN for each individual patient's age category.
8. Adequate biological parameters:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L
   2. Platelet count ≥100,000/mm3 (100 × 109/L)
   3. Hemoglobin ≥9 g/dL.
   4. Adequate immunoglobulin levels (IgG, IgA, IgM) that, in the opinion of the investigator, will not place the patient at increased risk for infection.
   5. Serum amylase and lipase <2 x ULN.
   6. Non-fasting serum triglyceride ≤300 mg/dL and non-fasting serum cholesterol ≤300 mg/dL, collected within 1 to 4 hours following a meal.
9. If receiving prescribed medication to prevent or treat seizures, the patient must be receiving stable doses for at least 1 month prior to screening visit.
10. Sexually active males with female partners of child-bearing potential or non-pregnant and non-breast feeding female of child-bearing potential:

    * Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting IP throughout 3 months after last dose of IP and have a negative urine pregnancy test (β-hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if the patient has had a tubal ligation.
    * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after the last dose of IP. A second form of birth control is required even if the patient has undergone a successful vasectomy.
11. The patient (when applicable) or the patient's parent(s) or legal guardian(s) understand(s) and voluntarily signed the informed consent document(s) prior to any study-related assessments/procedures being conducted.
12. The patient or parent(s)/guardian(s) is/are willing and able to comply with the study visit schedule and other protocol requirements, in the opinion of the investigator.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply at screening:

1. Renal insufficiency that, in the opinion of the investigator, requires or may require dialysis during the treatment and follow-up periods.
2. Cardiac ejection fraction/shortening fraction ≤50 % and/or severe end-organ hypo-perfusion syndrome (secondary to cardiac failure) resulting in lactic acidosis.
3. Patients with implanted cardiac assist/medical devices (including pacemakers), unless device was implanted prophylactically, and the patient is clinically asymptomatic.
4. In the opinion of the investigator, clinically significant ECG and/or ECHO findings at the time of screening.
5. Myocardial infarction within 6 months prior to enrollment.
6. Symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or unstable coronary artery disease.
7. Prior exposure to ABI-009, sirolimus, everolimus, or any other known rapamycin derivative, or previous treatment with any known mTOR inhibitor.
8. Patients who are breast feeding or have a confirmed or suspected pregnancy.
9. Treatment with any investigational drug (ie, a drug for which there is no approved indication), including an investigational drug for mitochondrial disease within 1 month prior to receiving the first dose of study drug (or within 3 months for a trial with an investigational biologic).
10. Disease-related surgical intervention within 1 month prior to the first dose of study drug.
11. Use of supplements that are contraindicated in the opinion of investigator, including super-fortified foods and/or beverages that include coenzyme Q10, Vitamin C, Vitamin E, and/or idebenone, etc, unless receiving stable doses for a minimum of 30 days prior to enrollment. Changes to mitochondrial dietary supplements or their doses for 30 days prior to enrollment.
12. Known hypersensitivity to ABI-009 (nab-sirolimus; ie, sirolimus and albumin), to any of its excipients, or to any known rapamycin derivative or known mTOR inhibitor.
13. Patients with confirmed or suspected increased intracranial pressure, pseudotumor cerebri (PTC)/idiopathic intracranial hypertension, and/or papilledema.
14. Any uncontrolled serious illness or psychiatric condition, medical condition, or other medical history, including abnormal laboratory test results which, in the opinion of the investigator, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results of the study.
15. Currently active malignancy (other than adequately treated non-melanoma skin cancers [ie, squamous cell and/or basal cell carcinoma], carcinoma in situ of the cervix, or other adequately treated carcinoma in situ) and/or ongoing treatment for malignancy are ineligible. Patients are not considered to have a currently active malignancy if they have completed therapy and are free of disease for ≥1 year.
16. Recent infection requiring systemic anti-infective treatment that was completed ≤14 days prior to enrollment.
17. Confirmed or suspected immunodeficiency disorder(s), including but not limited to, common variable immune deficiency (CVID), complement deficiency, etc.
18. Uncontrolled diabetes mellitus, as defined by HbA1c >8%, despite adequate therapy.
19. History of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
20. Use of strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4 (CYP3A4) and/or p-glycoprotein (p-GP) within the 14 days prior to receiving the first dose of study drug. Additionally, use of any known CYP3A4 substrates with a narrow therapeutic window (eg, fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfenadine) within the 14 days prior to receiving the first dose of study drug. [All medications will be reviewed by the (Institutional) Investigational Pharmacy to ensure that strong inducers and/or inhibitors of CYP3A4 and/or p-GP, or CYP3A4 substrates with a narrow therapeutic window, have not been administered within 14 days prior to the first dose of study drug; patients receiving anticonvulsant medications within the 14 days prior to receiving the first dose of study drug may be enrolled at the discretion of the investigator].
21. Known human immunodeficiency virus (HIV), active hepatitis B or hepatitis C infection(s).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events in pediatric patients with genetically-confirmed Leigh or Leigh-like syndrome administered ABI-009 intravenously (IV) | Up to 24 weeks
  Adverse events will be measured according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.